CLINICAL TRIAL: NCT06916130
Title: A Randomized, Open-label, Multiple Oral-dose, 2x2 Crossover Clinical Trial to Compare the Safety, Pharmacokinetic, and Pharmacodynamic Characteristics of a AD-120 and AD-120A in Healthy Adult Volunteers
Brief Title: A Study to Compare PK/PD Characteristics and Safety Profiles Between AD-120 and AD-120A
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-120PK/PD
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm-A (Experimental): Period 1 : Test Drug (AD-120), Period 2 : Reference Drug (AD-120A)
  Interventions: Drug: AD-120A; Drug: AD-120
- Arm-B (Experimental): Period 1 : Reference Drug (AD-120A), Period 2 : Test Drug (AD-120)
  Interventions: Drug: AD-120A; Drug: AD-120

INTERVENTIONS:
Drug: AD-120A — Administered before the breakfast during 7 days, Oral, Tablet
  Other Names: Reference Drug
Drug: AD-120 — Administered before the breakfast during 7 days, Oral, Tablet
  Other Names: Test drug

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic and pharmacodynamic characteristics of AD-120 in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic and pharmacodynamic characteristics and safety profiles of AD-120 compared with AD-120A in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50.0kg and equal to or less than 90.0kg and Body mass index (BMI) between 18.5 kg/m2 and 29.9 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 and equal to or less than 50 in healthy volunteers at the time of screening visit
* Negative result from Serum Helicobacter pylori antibody at the time of screening visit

Exclusion Criteria:

* Patients with trouble performing pH monitor catheter

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve over a dosing interval at steady state (AUCτ,ss) | AUCτ,ss: pre-dose to 24 hours of 1st administration versus pre-dose to 24 hours of repeated administration (7days)
  AUCτ,ss after 7days repeated administration of Omeprazole
The time of peak concentration after single dose | Tmax: from pre-dose to 24 hours of 1st administration
  Tmax after 1days administration of Omeprazole
Percent decrease from baseline in integrated gastric acidity measured by 24h pH monitoring | 24 hours before 1st administration to 24 hours after repeated administration (7days)
  Percent decrease from baseline in integrated gastric acidity measured by 24h pH monitoring for 24-hour interval after 7th dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea